CLINICAL TRIAL: NCT04067752
Title: Nutrition, Inflammation and Insulin Resistance in End-Stage Renal Disease
Acronym: SummerMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEPH-010-18F
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: End-stage Renal Disease
Keywords: dialysis; ESRD; hemodialysis; MRI
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: The design is randomized, cross-over, double-blind, placebo-controlled. Once the subject is determined to be eligible for the study, we will randomly assign him/her to one of the study arms (Dialysate Na concentration 138 mEq/L versus 132 mEq/L)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients will be randomized by computer generated sequence and study coordinators and co-investigators other than the primary investigator will be unblended to the treatment arms.
  The data will be sent to biostatistician with no identifiable information regarding randomization arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Dialysate Na (Experimental): high dialysate sodium concentration (138 mEq/L)
  Interventions: Other: high dialysate sodium concentration (138 mEq/L)
- Low Dialysate Na (Active Comparator): Low dialysate sodium concentration (132 mEq/L)
  Interventions: Other: Low dialysate sodium concentration

INTERVENTIONS:
Other: high dialysate sodium concentration (138 mEq/L) — high dialysate sodium concentration (138 mEq/L)
  Arms: High Dialysate Na
Other: Low dialysate sodium concentration — low dialysate sodium concentration (132 mEq/L)
  Arms: Low Dialysate Na

SUMMARY:
By 2030 an estimated 2 million people in the US will need dialysis or transplantation. Insulin resistance and chronic inflammation are common in dialysis patients and have been linked to protein-energy wasting, the most important determinant of clinical outcome in this patient population. The investigators hypothesize that the skin and muscle tissue sodium accumulation is a critical mechanism by which chronic inflammatory response and insulin resistance, alone or in combination lead to protein energy wasting in hemodialysis patients. The investigators will test this hypothesis by studying dialysis patients and matched controls without kidney disease by examining tissue Na content, markers of inflammation and protein metabolism.

DETAILED DESCRIPTION:
There are more than 420,000 patients receiving maintenance hemodialysis therapy in the United States, which is estimated to rise to over 500,000 patients by 2020. There are an estimated 45,500 Veterans receiving hemodialysis, of which over 3,000 enrolled Veterans were receiving dialysis at VA facilities in FY 2013. Over the last decade, there have been no therapies proven to significantly lower the mortality and morbidity risk for these patients. One of the most important determinants of this poor clinical outcome is protein energy wasting, a highly prevalent nutritional and metabolic abnormality characterized by increased protein breakdown in the skeletal muscle compartment. The investigators' group has shown that two well-recognized and interrelated metabolic abnormalities, insulin resistance and persistent inflammation, are likely to play a critical role in the pathogenesis of protein energy wasting and related nutritional and metabolic abnormalities. The investigators' preliminary data show that in maintenance hemodialysis (MHD) patients 1) There is an inadequate response to protein anabolic actions of insulin; 2) Persistent systemic inflammation is strongly and independently associated with skeletal muscle net protein balance; and 3) Pharmacological modulation of systemic inflammation and insulin resistance partially, but not fully, reverse net protein catabolism. It was demonstrated that non-osmotic sodium (Na) is stored in skin and muscle without commensurate water retention, which leads to local immune-cell activation and accelerated pro-inflammatory status. The investigators' preliminary data show that the skin and muscle Na+ contents, derived by 23Na magnetic resonance imaging (MRI) are substantially higher in MHD patients compared to matched healthy controls. The investigators also showed that increased skin and muscle Na concentrations are significantly associated with increased inflammatory response and decreased peripheral insulin sensitivity, in patients on MHD. These data suggest that tissue Na content, immune pathways and insulin resistance are closely linked and could lead to increased risk for protein energy wasting in MHD patients. It was reported that standard 4-hour conventional hemodialysis provides significant Na removal from muscle and skin suggesting that tissue Na and water content could be modulated by modulating hemodialysis prescription. The overall goal of this application is to elucidate the mechanisms by which tissue sodium accumulation, persistent immune system activation and insulin resistance influence the development of protein energy wasting in MHD patients. The investigators hypothesize that the skin and muscle tissue sodium accumulation is a critical mechanism by which chronic inflammatory response and insulin resistance, alone or in combination, lead to protein energy wasting in MHD patients. Specific Aims: To test the hypothesis that removal of tissue sodium by modulating hemodialysis prescription would improve metabolic milieu and protein energy wasting in MHD patients. The investigators will achieve this goal through a cross-over randomized clinical trial whereby dialysate sodium concentrations will be modulated (138 mEq/L versus 132 mEq/L, 4 weeks each) to remove 10% of baseline skeletal muscle Na content in the setting of stable sodium intake by diet. The primary outcomes will be markers of net protein balance, inflammation, and macronutrient disposal rates. If successful, the proposed studies will have great potential to influence clinical practices in MHD patients because the proposed intervention protocol would be easily accessible and could ultimately lead to improvements in the hospitalization and death rates with great impact on Veterans' Health Care and make important contributions to the research mission of the Department of Veterans Administration.

ELIGIBILITY:
Inclusion Criteria:

* On MHD for more than 6 months
* Have acceptable dialysis adequacy (eKt/V > 1.2) for a minimum of 3 months and a patent, well-functioning, hemodialysis AV access
* Ability to give informed consent

Exclusion Criteria:

* Pregnancy
* Intolerance to the medication in metabolic studies)
* Presence of a metal object in the body that might interfere with MRI
* Severe, unstable, active, or chronic inflammatory disease (active infection, active connective tissue disorder, active cancer or cancer history in the prior 5 years, HIV, liver disease, active chronic hepatitis B or C)
* Type 1 Diabetes on insulin therapy; Hospitalization within 1 month prior to the study
* Receiving steroids (including inhaled steroid and high potency topical, with the exception of over the counter hydrocortisone cream
* Prednisone > 5 mg/day) and/or other immunosuppressive agents
* Residual renal function > 5ml/min or urine output > 400 ml/day

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Net whole-body muscle protein balance measured by stable isotope technique reported as mg/kg.fat free mass/min | 4 weeks
  Net whole-body muscle protein balance measured by stable isotope technique reported as mg/kg.fat free mass/min. This reflects the balance between endogenous leucine appearance rate (protein synthesis), the leucine oxidation rate, and the non-oxidative leucine disappearance rate (protein breakdown).
Net skeletal muscle protein balance measured by stable isotope technique reported as g/100 ml/min | 4 weeks
  Net skeletal muscle protein balance measured by stable isotope technique reported as g/100 ml/min. This reflects the dilution and enrichment of phenylalanine across the forearm. Because phenylalanine is neither synthesized nor metabolized by skeletal muscle, rate of appearance (Ra) of unlabeled phenylalanine reflects muscle protein breakdown, whereas the rate of disappearance (Rd) of labeled phenylalanine estimates muscle protein synthesis. the difference between synthesis and breakdown provides net skeletal muscle protein balance at a given rate of blood flow.
Muscle sodium content | 4 weeks
  Muscle sodoium content measured by NAMRI before and after intervention
Skin sodium content | 4 weeks
  Skin sodium content measured by NAMRI before and after intervention

SECONDARY OUTCOMES:
Handgrip strength measured by dynamometer | 4 weeks
  Handgrip strength (HGS) will be measured on the non stula side before dialysis session using a Jamar hydraulic dynamometer.
Recovery time | 4 weeks
  Patients will be asked how long it took them to recover completely from the preceding session
Pulse Wave Velocity | 4 weeks
  Pulse Wave Velocity will be measured by Sphygmocor.
Interleukin 6 | 4 weeks
  proinflammatory cytokine IL6 will be measured as a inflammatory marker
Sit to stand test | 4 weeks
  measurement of how many sit to stands can be accomplished at a given time period to assess physical function
Short Physical Performance Battery | 4 weeks
  Balance, gait speed and chair speed tests will be scored to provide a complete score to assess physical function
6-minute walk | 4 weeks
  measurement of how long can a patient walk within 6 minutes to assess physical function
hsCRP | 4 weeks
  hsCRP will be measured as a marker of systemic inflammation
Interleukin 1 | 4 weeks
  Proinflammatory cytokine Interleukin 1 (IL1) will be measured as a inflammatory marker

CONTACTS AND LOCATIONS:
Overall Officials: Talat A Ikizler, MD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (2):
- United States (2):
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Vanderbilt University Medical center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ertuglu LA, Sahinoz M, Alsouqi A, Deger SM, Guide A, Pike M, Robinson-Cohen C, Akwo E, Pridmore M, Crescenzi R, Madhur MS, Kirabo A, Harrison DG, Luft FC, Titze J, Ikizler TA, Gamboa JL. Intermuscular adipose tissue accumulation is associated with higher tissue sodium in healthy individuals. Physiol Rep. 2024 Jul;12(13):e16127. doi: 10.14814/phy2.16127. PMID 38960895

DOCUMENTS (1):
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT04067752/ICF_000.pdf